CLINICAL TRIAL: NCT03571425
Title: The Impact of Enteral Versus Oral Protein Feeding on Muscle Protein Synthesis in Healthy Young Males and Females
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Exeter (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 180509/B/03
Record Dates: First submitted 2018-05-24; First posted 2018-06-27 (Actual); Last update posted 2018-12-20 (Actual); Status verified 2018-12

CONDITIONS: Healthy
MeSH Terms: interventions — Proteins

STUDY DESIGN:
Masking Description: Oral conditions are double blinded to participant and investigator, but enteral vs oral feeding is not blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (3):
- Oral Placebo (Placebo Comparator): Placebo drink
  Interventions: Other: Oral Placebo
- Oral Protein (Active Comparator): Protein drink, ingested orally
  Interventions: Other: Oral Protein
- Enteral Protein (Active Comparator): Protein drink, administered via enteral tube
  Interventions: Other: Enteral Protein

INTERVENTIONS:
Other: Oral Placebo — A placebo beverage will be consumed orally
  Arms: Oral Placebo
Other: Oral Protein — A protein beverage will be consumed orally
  Arms: Oral Protein
Other: Enteral Protein — A protein beverage will be consumed via a naso-gastric feeding tube
  Arms: Enteral Protein

SUMMARY:
The present study will seek to quantify the muscle protein synthetic response to a protein beverage consumed orally or through a nasogastric tube in healthy, young individuals.

DETAILED DESCRIPTION:
Thirty healthy, young volunteers will receive a stable isotope tracer infusion (8.5h) combined with repeated blood and muscle sampling, in order to measure muscle protein synthesis rate in the postabsorptive state, and following oral placebo ingestion (n=10), oral protein ingestion (n=10), or enteral protein administration (n=10).

ELIGIBILITY:
Inclusion Criteria:

* 18-40 years of age
* Body mass index between 18.5 and 30

Exclusion Criteria:

* Any diagnosed metabolic impairment (e.g. type 1 or 2 Diabetes)
* Any diagnosed cardiovascular disease
* Elevated blood pressure at the time of screening. (An average systolic blood pressure reading of ≥140 mmHg over two or more measurements and an average diastolic blood pressure of ≥90 mmHg over two or more measurements)
* Chronic use of any prescribed or over the counter pharmaceuticals (that may modulate muscle protein metabolism). This excludes oral contraceptives and contraceptive devices.
* A personal or family history of epilepsy, seizures or schizophrenia.
* Presence of an ulcer in the stomach or gut and/or strong history of indigestion
* Known pre-existing liver disease/condition
* Any known disorders in muscle metabolism
* Regular use of nutritional supplements
* Allergy to lidocaine
* Allergy to milk
* Current paracetamol use (i.e. use of paracetamol more than once a week)
* Pregnancy

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2018-06-04 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2018-12-01 (Actual)

PRIMARY OUTCOMES:
Postprandial muscle protein synthesis | 5 hours
  Muscle protein synthesis rate (FSR) following ingestion of a placebo or protein supplement

SECONDARY OUTCOMES:
Postabsorptive muscle protein synthesis | 2 hours
  Muscle protein synthesis rate (FSR, in %/h) during a 2 hour fasting period
Whole-body protein synthesis | 7 hours
  Whole-body protein synthesis, measured using a D5 phenylalanine and D2 tyrosine infusion (umol Phenylalanine/kg/h)
Whole-body protein breakdown | 7 hours
  Whole-body protein breakdown, measured using a D5 phenylalanine and D2 tyrosine infusion (umol Phenylalanine/kg/h)
Whole-body protein oxidation | 7 hours
  Whole-body protein oxidation, measured using a D5 phenylalanine and D2 tyrosine infusion (umol Phenylalanine/kg/h)
Whole-body protein net balance | 7 hours
  Whole-body protein net balance, measured using a D5 phenylalanine and D2 tyrosine infusion (umol Phenylalanine/kg/h)
Gastric emptying rate | 5 hours
  Gastric emptying rate following ingestion of a placebo or protein drink
Blood glucose concentration | 8.5 hours
  Blood glucose concentration in the postabsorptive and postprandial phase following placebo/protein ingestion
Serum insulin concentration | 8.5 hours
  Serum insulin concentration in the postabsorptive and postprandial phase following placebo/protein ingestion

CONTACTS AND LOCATIONS:
Overall Officials: Marlou Dirks, PhD, Principal Investigator — University of Exeter
Locations (1):
- University of Exeter, Exeter, Devon, United Kingdom

IPD SHARING:
Plan to Share IPD: No